CLINICAL TRIAL: NCT01198145
Title: Phase III, Randomized, Study of Sulfasalazine Versus Placebo in the Prevention of Acute Diarrhea in Patients Receiving Pelvic Radiation Therapy
Brief Title: Sulfasalazine in Preventing Acute Diarrhea in Patients With Cancer Who Are Undergoing Pelvic Radiation Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N08C9; NCI-2011-02602 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000684240 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-04

CONDITIONS: Diarrhea; Gastrointestinal Complications; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: diarrhea; gastrointestinal complications; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Diarrhea | interventions — Sulfasalazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: Sulfasalazine (Experimental): Patients receive oral sulfasalazine twice daily during radiotherapy and for 4 weeks after completion of radiotherapy.
  Interventions: Drug: sulfasalazine
- Arm II: Placebo (Placebo Comparator): Patients receive oral placebo twice daily during radiotherapy and for 4 weeks after completion of radiotherapy.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: sulfasalazine — Given orally
  Arms: Arm I: Sulfasalazine
Other: placebo — Given orally
  Arms: Arm II: Placebo

SUMMARY:
RATIONALE: Sulfasalazine may relieve diarrhea in patients with cancer who are undergoing pelvic radiation therapy.

PURPOSE: This randomized phase III trial is studying sulfasalazine to see how well it works in preventing acute diarrhea in patients with cancer who are undergoing pelvic radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether sulfasalazine is effective in reducing the acute treatment-related diarrhea in patients receiving pelvic radiotherapy as measured by NCI CTC v4.0 in patients receiving pelvic external-beam radiotherapy as adjuvant or primary treatment for malignancy.

Secondary

* To determine whether sulfasalazine can reduce chronic treatment-related bowel dysfunction following completion of therapy.
* To determine whether sulfasalazine causes any toxicity in this situation.

Tertiary

* To bank blood products for future studies, as part of ongoing research for NCCTG studies (Mayo Clinic Rochester only). (Translational)

OUTLINE: This is a multicenter study. Patients are stratified according to history of anterior resection of the rectum (yes vs no); total planned cumulative dosing, including boost fields of external-beam radiotherapy (4500-5350 cGy vs > 5350 cGy); and concurrent radiosensitizing fluorouracil, capecitabine, or oxaliplatin (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral sulfasalazine twice daily during radiotherapy* and for 4 weeks after completion of radiotherapy.
* Arm II: Patients receive oral placebo twice daily during radiotherapy* and for 4 weeks after completion of radiotherapy.

NOTE: *Patients must start study treatment by the third radiotherapy fraction.

Patients may undergo blood sample collection at baseline and then weekly during radiotherapy. All patients complete quality of life and bowel function questionnaires at baseline, weekly during radiotherapy, and at 6 weeks after completion of radiotherapy.

After completion of radiotherapy, patients are followed up at 6 weeks and at 12 and 24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer that supports the use of radiotherapy to the pelvis
* No current or prior metastases beyond pelvic regional lymph nodes
* Planning to receive a course of continuous definitive or adjuvant external-beam radiotherapy to a minimum dose of 4500 cGy with or without fluorouracil, capecitabine, or oxaliplatin
* Planned course of pelvic radiotherapy must fall within the following parameters:

  * Pelvis must be encompassed by the planned radiotherapy fields

    * Superior border may not lie superior to the L4-5 interspace and may not be inferior to the most inferior aspect of the sacroiliac joints
    * Portions of the rectum may have special blocking, depending upon disease site
  * Total planned dose to the central axis midplane (for AP-PA parallel opposed fields) or isocenter (for 3- or 4-field techniques) for the pelvic field must lie between 4500-5300 cGy (inclusive)*

    * Subsequent to completion of treatment to the pelvic field, a boost to primary tumor or tumor bed may be planned
  * Planned treatment is to be given 4-5 times per week on a one-treatment-per-day basis

    * Daily dose (specified at central axis midplane or at isocenter for multi-field techniques) must lie between 170-210 cGy (inclusive) per day*
* NOTE: *For institutions that do not use midplane or isocenter as the point for specification of dose, it will be necessary to determine the dose according to the methods specified above in order to determine patient eligibility.
* No perineal irradiation planned (e.g., anal cancer patients, patients who have had an abdominal-perineal resection)
* No brachytherapy planned before the completion of all external-beam radiotherapy
* No planned split-course radiotherapy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 6 months
* Hemoglobin ≥ 10.0 g/dL
* Leukocytes ≥ 3,500/mm^3
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* AST ≤ 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Willing to provide blood specimens as required by the study (Mayo Clinic Rochester patients only)
* Able to complete questionnaires alone or with assistance
* No history of inflammatory bowel disease
* No history of gastrointestinal or genitourinary obstruction or porphyria
* No history of G6PD deficiency
* No history of irritable bowel syndrome
* No history of blood dyscrasia
* No history of severe allergies or asthma
* No history of hepatic or renal disease
* No diarrhea ≥ grade 3, rectal bleeding, abdominal cramping, or incontinence of stool within the past week
* No medical condition that may interfere with the ability to receive study treatment
* No known allergy to sulfasalazine, sulfa medications, salicylates, or any known component of drug formulation

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior pelvic radiotherapy
* No prior abdominal-perineal resection, Hartmann procedure, or other surgical procedure leaving the patient without a functioning rectum
* No planned use of leucovorin or cytotoxic chemotherapeutic agents concurrent with radiotherapy (except for fluorouracil, capecitabine, or oxaliplatin)
* No other concurrent sulfasalazine
* No concurrent digoxin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2013-07-22 (Actual); Study Completion 2017-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Miller, MD, Study Chair — Mayo Clinic
Locations (257):
- United States (257):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - St. Francis Hospital Cancer Care Services, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Mercy Cancer Center - West Lakes, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Union Hospital of Cecil County, Elkton, Maryland
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - St. Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Duluth Clinic, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - Central Care Cancer Center at Carrie J. Babb Cancer Center, Bolivar, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Goldschmidt Cancer Center, Jefferson City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - University of New Mexico Cancer Center - South, Las Cruces, New Mexico
  - Mount Kisco Medical Group, PC, Mount Kisco, New York
  - Randolph Hospital, Asheboro, North Carolina
  - CaroMont Cancer Center at Gaston Memorial Hospital, Gastonia, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Park Ridge Hospital, Hendersonville, North Carolina
  - High Point Regional Hospital, High Point, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - AnMed Cancer Center, Anderson, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Ravenel Oncology Center at Memorial Hospital of Martinsville and Henry County, Martinsville, Virginia
  - Legacy Salmon Creek Medical Center, Vancouver, Washington
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - Center for Cancer Treatment & Prevention at Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Central Wisconsin Cancer Program at Agnesian HealthCare, Fond du Lac, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital Cancer Center, Stevens Point, Wisconsin
  - Door County Cancer Center at Door County Memorial Hospital, Sturgeon Bay, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Ministry Saint Clare's Hospital, Weston, Wisconsin

REFERENCES:
- [Derived] Miller RC, Petereit DG, Sloan JA, Liu H, Martenson JA, Bearden JD 3rd, Sapiente R, Seeger GR, Mowat RB, Liem B, Iott MJ, Loprinzi CL; Alliance for Clinical Trials in Oncology. N08C9 (Alliance): A Phase 3 Randomized Study of Sulfasalazine Versus Placebo in the Prevention of Acute Diarrhea in Patients Receiving Pelvic Radiation Therapy. Int J Radiat Oncol Biol Phys. 2016 Jul 15;95(4):1168-74. doi: 10.1016/j.ijrobp.2016.01.063. Epub 2016 Apr 23. PMID 27354129
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: Sulfasalazine: Patients receive two 500 mg oral sulfasalazine tablets twice daily during radiotherapy and for 4 weeks after completion of radiotherapy.
- Arm II: Placebo: Patients receive two oral placebo tablets twice daily during radiotherapy and for 4 weeks after completion of radiotherapy.
  >
  > placebo: Given orally
Period: Overall Study
Arm/Group | Arm I: Sulfasalazine | Arm II: Placebo
Started | 44 | 43
Completed | 43 | 42
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Two patients in Arm I and one patient from Arm II were not included in the baseline analysis nor the endpoint analyses due to cancellations and protocol violations.
Groups:
- Arm II: Placebo: Patients receive two oral placebo tablets twice daily during radiotherapy and for 4 weeks after completion of radiotherapy.>
  > placebo: Given orally
- Total: Total of all reporting groups
Arm/Group | Arm I: Sulfasalazine | Arm II: Placebo | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Continuous [Median (Full Range); unit: years] | 59 [37 to 84] | 56.5 [37 to 81] | 58 [37 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 33
  Male | 27 | 24 | 51
Region of Enrollment [Number; unit: participants]
  United States | 42 | 42 | 84

OUTCOME MEASURES:

1. Primary Outcome: Maximum Severity of Diarrhea Toxicity as Measured by the CTCAE v4.0 During and After Radiotherapy (RT)
Description: The primary endpoint for this study is the maximal severity of diarrhea toxicity. Severity of diarrhea was graded using the terminology and grading categories defined in the NCI's Common Toxicity Criteria (CTCAE), Version 4.0. Grade 0 = None; 1=Mild; Grade 2=Moderate, Grade 3=Severe, Grade 4=Life-threatening as measured by the CTCAE version 4.0. Assessments were recorded during the course of RT and for 6 weeks following RT. The table below represents the worst graded diarrhea for each patient.
  A two-sided Wilcoxon rank-sum test will be used to test the equality of the distributions of maximum diarrhea severity grades between the two treatment arms.
Time Frame: During radiation therapy and up to 6 weeks post radiation therapy
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I: Sulfasalazine | Arm II: Placebo
Number analyzed (Participants) | 42 | 42
Participants
  Grade 0 | 10 | 10
  Grade 1 | 13 | 15
  Grade 2 | 8 | 13
  Grade 3 | 10 | 4
  Grade 4 | 1 | 0
Statistical Analysis 1: Comparison: Arm I: Sulfasalazine vs Arm II: Placebo; Test type: Superiority or Other; p = 0.41, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Maximum Severity of Each Outcome Variable (Rectal Bleeding, Abdominal Cramping, Tenesmus, Constipation, and Diarrhea) Measured During and After RT
Description: The maximal severity of each of 5 different adverse even types (Tenesmus, Abdominal Pain, Constipation, Diarrhea, and Rectal Bleeding) were collected as a secondary endpoint. Severity of the events was graded using the terminology and grading categories defined in the NCI's Common Toxicity Criteria (CTCAE), Version 4.0. Grade 0 = None; 1=Mild; Grade 2=Moderate, Grade 3=Severe, Grade 4=Life-threatening. Adverse events were assessed during the course of RT and for 6 weeks following RT. The table below represents the worst grade for each patient for each type.
  Two-sided chi-square tests will be used to compare each percentage variable between treatment arms for each event type.
Time Frame: During radiation therapy and up to 6 weeks post radiation therapy
Population: Two patients in Arm I and one patient from Arm II were not included in the endpoint analyses due to cancellations and protocol violations. 42 patients from each arm started RT and were used for the analysis. 25 patients from Arm I and 29 patients from Arm II were evaluated after RT. Two patients from Arm 1 provided incomplete data.
Measure: Count of Participants; unit: Participants
Groups:
- Arm II: Placebo: Patients receive two oral placebo tablets twice daily during radiotherapy and for 4 weeks after completion of radiotherapy.
Arm/Group | Arm I: Sulfasalazine | Arm II: Placebo
Number analyzed (Participants) | 42 | 42
Participants
  Tenesmus during RT: Grade 0 | 27 | 30
  Tenesmus during RT: Grade 1 | 6 | 9
  Tenesmus during RT: Grade 2 | 7 | 3
  Tenesmus during RT: Grade 3 | 2 | 0
  Tenesmus during RT: Grade 4 | 0 | 0
  Tenesmus after RT: number analyzed (Participants) | 23 | 29
  Tenesmus after RT: Grade 0 | 18 | 21
  Tenesmus after RT: Grade 1 | 5 | 7
  Tenesmus after RT: Grade 2 | 0 | 1
  Tenesmus after RT: Grade 3 | 0 | 0
  Tenesmus after RT: Grade 4 | 0 | 0
  Abdominal pain during RT: Grade 0 | 22 | 26
  Abdominal pain during RT: Grade 1 | 14 | 12
  Abdominal pain during RT: Grade 2 | 3 | 4
  Abdominal pain during RT: Grade 3 | 3 | 0
  Abdominal pain during RT: Grade 4 | 0 | 0
  Abdominal pain after RT: number analyzed (Participants) | 25 | 29
  Abdominal pain after RT: Grade 0 | 17 | 24
  Abdominal pain after RT: Grade 1 | 8 | 2
  Abdominal pain after RT: Grade 2 | 0 | 3
  Abdominal pain after RT: Grade 3 | 0 | 0
  Abdominal pain after RT: Grade 4 | 0 | 0
  Constipation during RT: Grade 0 | 26 | 27
  Constipation during RT: Grade 1 | 12 | 13
  Constipation during RT: Grade 2 | 4 | 2
  Constipation during RT: Grade 3 | 0 | 0
  Constipation during RT: Grade 4 | 0 | 0
  Constipation after RT: number analyzed (Participants) | 25 | 29
  Constipation after RT: Grade 0 | 19 | 22
  Constipation after RT: Grade 1 | 6 | 6
  Constipation after RT: Grade 2 | 0 | 1
  Constipation after RT: Grade 3 | 0 | 0
  Constipation after RT: Grade 4 | 0 | 0
  Diarrhea during RT: Grade 0 | 10 | 11
  Diarrhea during RT: Grade 1 | 13 | 14
  Diarrhea during RT: Grade 2 | 9 | 13
  Diarrhea during RT: Grade 3 | 9 | 4
  Diarrhea during RT: Grade 4 | 1 | 0
  Diarrhea after RT: number analyzed (Participants) | 25 | 29
  Diarrhea after RT: Grade 0 | 11 | 14
  Diarrhea after RT: Grade 1 | 12 | 10
  Diarrhea after RT: Grade 2 | 2 | 3
  Diarrhea after RT: Grade 3 | 0 | 2
  Diarrhea after RT: Grade 4 | 0 | 0
  Rectal bleeding during RT: Grade 0 | 26 | 22
  Rectal bleeding during RT: Grade 1 | 16 | 20
  Rectal bleeding during RT: Grade 2 | 0 | 0
  Rectal bleeding during RT: Grade 3 | 0 | 0
  Rectal bleeding during RT: Grade 4 | 0 | 0
  Rectal bleeding after RT: number analyzed (Participants) | 25 | 29
  Rectal bleeding after RT: Grade 0 | 20 | 27
  Rectal bleeding after RT: Grade 1 | 5 | 2
  Rectal bleeding after RT: Grade 2 | 0 | 0
  Rectal bleeding after RT: Grade 3 | 0 | 0
  Rectal bleeding after RT: Grade 4 | 0 | 0
Statistical Analysis 1: Comparison: Arm I: Sulfasalazine vs Arm II: Placebo; Comparing Tenesmus During RT; Test type: Superiority or Other; p = 0.23, Chi-squared
Statistical Analysis 2: Comparison: Arm I: Sulfasalazine vs Arm II: Placebo; Comparing Tenesmus after RT; Test type: Superiority or Other; p = 0.64, Chi-squared
Statistical Analysis 3: Comparison: Arm I: Sulfasalazine vs Arm II: Placebo; Comparing abdominal pain during RT; Test type: Superiority or Other; p = 0.30, Chi-squared
Statistical Analysis 4: Comparison: Arm I: Sulfasalazine vs Arm II: Placebo; Comparing abdominal pain after RT; Test type: Superiority or Other; p = 0.02, Chi-squared
Statistical Analysis 5: Comparison: Arm I: Sulfasalazine vs Arm II: Placebo; Comparing constipation during RT; Test type: Superiority or Other; p = 0.70, Chi-squared
Statistical Analysis 6: Comparison: Arm I: Sulfasalazine vs Arm II: Placebo; Comparing constipation after RT; Test type: Superiority or Other; p = 0.63, Chi-squared
Statistical Analysis 7: Comparison: Arm I: Sulfasalazine vs Arm II: Placebo; Comparing diarrhea during RT; Test type: Superiority or Other; p = 0.44, Chi-squared
Statistical Analysis 8: Comparison: Arm I: Sulfasalazine vs Arm II: Placebo; Comparing diarrhea after RT; Test type: Superiority or Other; p = 0.48, Chi-squared
Statistical Analysis 9: Comparison: Arm I: Sulfasalazine vs Arm II: Placebo; Comparing rectal bleeding during RT; Test type: Superiority or Other; p = 0.38, Chi-squared
Statistical Analysis 10: Comparison: Arm I: Sulfasalazine vs Arm II: Placebo; Test type: Superiority or Other; p = 0.15, Chi-squared

3. Secondary Outcome: Area Under the Curve That Combines the Individual Severity of Diarrhea Toxicity as Measured by the CTCAE v4.0 During and After RT
Description: For each patient, an Area Under the Curve (AUC) summary statistic will be calculated taking into account the individual severity of diarrhea toxicity over time. Severity of diarrhea was graded using the terminology and grading categories defined in the NCI's Common Toxicity Criteria (CTCAE), Version 4.0. Grade 0 = None; 1=Mild; Grade 2=Moderate, Grade 3=Severe, Grade 4=Life-threatening. The curve was constructed using weekly assessments during and after RT. A separate analysis was done during the course of RT and every week for 6 weeks following RT.
Time Frame: During radiation therapy and up to 6 weeks post radiation therapy
Population: Two patients in Arm I and one patient from Arm II were not included in the endpoint analyses due to cancellations and protocol violations. 42 patients from each arm started RT and were used in that portion of the analysis. 25 patients from Arm I and 29 patients from Arm II were evaluated after RT. Two patients from Arm 1 provided incomplete data.
Measure: Mean (Standard Deviation); unit: grade*week
Arm/Group | Arm I: Sulfasalazine | Arm II: Placebo
Number analyzed (Participants) | 42 | 42
grade*week
  During RT | 4.0 (3.9) | 3.3 (3.0)
  After RT: number analyzed (Participants) | 29 | 25
  After RT | 1.2 (1.7) | 1.3 (2.4)
Statistical Analysis 1: Comparison: Arm I: Sulfasalazine vs Arm II: Placebo; Result comparing Arm I and Arm II during RT; Test type: Superiority or Other; p = 0.56, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm I: Sulfasalazine vs Arm II: Placebo; Result comparing Arm I and Arm II after RT; Test type: Superiority or Other; p = 0.74, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Average Graded Severity for Tenesmus, Abdominal Pain, Constipation, Diarrhea and Hemorrhage During and After RT as Graded by CTCAE v4.0
Description: Tenesmus, Abdominal pain, constipation, diarrhea and hemorrhaging were assessed during RT and up to 6 weeks after RT. Severity of these events were graded using the terminology and grading categories defined in the NCI's Common Toxicity Criteria (CTCAE), Version 4.0. Grade 0 = None; 1=Mild; Grade 2=Moderate, Grade 3=Severe, Grade 4=Life-threatening. For each patient, an average score for each outcome variable during and after RT calculated as follows: The sum of all severity scores for that variable divided by the number of severity scores for that variable recorded for the patient during the course of RT and for 6 weeks following RT.
Time Frame: During radiation therapy and up to 6 weeks post radiation therapy
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Average Grade of Event
Arm/Group | Arm I: Sulfasalazine | Arm II: Placebo
Number analyzed (Participants) | 42 | 42
Average Grade of Event
  Tenesmus during RT | 0.2 (0.4) | 0.1 (0.2)
  Tenesmus after RT: number analyzed (Participants) | 23 | 29
  Tenesmus after RT | 0.1 (0.2) | 0.1 (0.4)
  Abdominal pain during RT | 0.3 (0.4) | 0.2 (0.3)
  Abdominal pain after RT: number analyzed (Participants) | 25 | 29
  Abdominal pain after RT | 0.2 (0.3) | 0.2 (0.4)
  Constipation during RT | 0.2 (0.3) | 0.2 (0.3)
  Constipation after RT: number analyzed (Participants) | 25 | 29
  Constipation after RT | 0.1 (0.3) | 0.1 (0.2)
  Diarrhea during RT | 0.8 (0.7) | 0.6 (0.6)
  Diarrhea after RT: number analyzed (Participants) | 25 | 29
  Diarrhea after RT | 0.3 (0.4) | 0.3 (0.4)
  Rectal bleeding during RT | 0.2 (0.3) | 0.2 (0.3)
  Rectal bleeding after RT: number analyzed (Participants) | 25 | 29
  Rectal bleeding after RT | 0.1 (0.3) | 0.1 (0.2)

5. Secondary Outcome: Percentage of Patients in Each Arm That Experience Tenesmus, Abdominal Pain, Constipation, Diarrhea and Rectal Bleeding During and After RT
Description: The number of patients that reported any grade 1 or higher adverse event was divided by the total number of patients evaluated. The analysis was done separately for each of the 5 outcomes and separately during RT and after RT.
Time Frame: During radiation therapy and up to 6 weeks post radiation therapy
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Arm I: Sulfasalazine | Arm II: Placebo
Number analyzed (Participants) | 42 | 42
percentage of participants
  Tenesmus during RT | 35.7 | 28.6
  Tenesmus after RT: number analyzed (Participants) | 23 | 29
  Tenesmus after RT | 11.9 | 19.1
  Abdominal pain during RT | 47.6 | 38.1
  Abdominal pain after RT: number analyzed (Participants) | 25 | 29
  Abdominal pain after RT | 19.1 | 11.9
  Constipation during RT | 38.1 | 35.7
  Constipation after RT: number analyzed (Participants) | 25 | 29
  Constipation after RT | 14.3 | 16.7
  Diarrhea during RT | 76.2 | 73.8
  Diarrhea after RT: number analyzed (Participants) | 25 | 29
  Diarrhea after RT | 33.3 | 35.7
  Rectal bleeding during RT | 38.1 | 47.6
  Rectal bleeding after RT: number analyzed (Participants) | 25 | 29
  Rectal bleeding after RT | 11.9 | 4.8

6. Secondary Outcome: Percent of Patients in Each Arm That Recorded "Yes" to Each of Questions 2-10 on the Bowel Function Questionnaire
Description: Questions that were used in this analysis:
  2. Have you had a problem causing you to get up at night to have a bowel movement? 3. Have you had a problem causing you to lose control of your bowel movements? 4. Have you had a problem causing you to have a bowel movement within 30 minutes of a prior bowel movement? 5. Have you had to wear protective clothing or a pad in case you lost control of a bowel movement? 6. Have you had a problem causing you to be unable to tell the difference between stool and gas? 7. Have you had a problem causing you to have stools that are liquid? 1=yes 2=no q08 8. Have you found that once you feel the urge to have a bowel movement, you must do so within 15 minutes to avoid an accident? 9. Have you had cramping with a bowel movement? 10. Have you had blood in your bowel movement?
Time Frame: Up to 6 weeks post radiation therapy
Population: All patients that completed the questionnaire were included in the analysis. Questionnaires used were completed during the last week during RT and 6 weeks after RT.
Measure: Number; unit: percentage of participants
Arm/Group | Arm I: Sulfasalazine | Arm II: Placebo
Number analyzed (Participants) | 39 | 41
percentage of participants
  During RT : Q2: number analyzed (Participants) | 28 | 32
  During RT : Q2 | 19 | 10
  During RT : Q3: number analyzed (Participants) | 28 | 32
  During RT : Q3 | 11 | 10
  During RT : Q4: number analyzed (Participants) | 28 | 32
  During RT : Q4 | 33 | 33
  During RT : Q5: number analyzed (Participants) | 28 | 32
  During RT : Q5 | 7 | 0
  During RT : Q6: number analyzed (Participants) | 28 | 32
  During RT : Q6 | 26 | 23
  During RT : Q7: number analyzed (Participants) | 28 | 32
  During RT : Q7 | 11 | 20
  During RT : Q8: number analyzed (Participants) | 28 | 32
  During RT : Q8 | 44 | 43
  During RT : Q9: number analyzed (Participants) | 28 | 32
  During RT : Q9 | 4 | 17
  During RT : Q10: number analyzed (Participants) | 28 | 32
  During RT : Q10 | 7 | 7
  After RT : Q2 | 39 | 27
  After RT : Q3 | 24 | 22
  After RT : Q4 | 55 | 56
  After RT : Q5 | 18 | 12
  After RT : Q6 | 37 | 46
  After RT : Q7 | 37 | 37
  After RT : Q8 | 70 | 61
  After RT : Q9 | 34 | 34
  After RT : Q10 | 50 | 29

7. Secondary Outcome: Percentage of Patients in Each Arm That Require Any Type of Antidiarrheal Medications.
Description: The number of patients reporting the use of anti-diarrheal medications divided by the number of patients evaluated for this endpoint.
Time Frame: Up to 24 months post radiotherapy
Population: Two patients in Arm I and one patient from Arm II were not included in the endpoint analyses due to cancellations and protocol violations.
Measure: Number; unit: percentage of participants
Arm/Group | Arm I: Sulfasalazine | Arm II: Placebo
Number analyzed (Participants) | 42 | 42
percentage of participants | 48.7 | 28.6

8. Secondary Outcome: Percentage of Patients in Each Arm That Experience Clinically Significant Deficits in Overall Quality of Life and Fatigue
Description: For each arm, the percentage of patients experience clinically significant deficits in overall QOL and fatigue as indicated by a score of 5 or lower on the 0-10 scale. The analysis was done using the questionnaire that was completed during the first week of radiotherapy (RT) and 6 weeks after RT.
Time Frame: Up to 6 weeks post radiotherapy
Population: All completed QOL questionnaires were included in the analysis. Questionnaires used were completed during the first week during RT and 6 weeks after RT. From Arm I, 41 patients completed questionnaires, 39 during and 26 after RT. For Arm II, 42 patients completed the questions, 40 during and 29 after RT.
Measure: Number; unit: percentage of participants
Arm/Group | Arm I: Sulfasalazine | Arm II: Placebo
Number analyzed (Participants) | 41 | 42
percentage of participants
  During RT: number analyzed (Participants) | 39 | 40
  During RT | 17.9 | 7.5
  After RT: number analyzed (Participants) | 26 | 29
  After RT | 26.9 | 27.6

ADVERSE EVENTS:
Arm/Group | Arm I: Sulfasalazine | Arm II: Placebo
Serious Adverse Events (participants affected / at risk) | 1/43 | 2/42
Other Adverse Events (participants affected / at risk) | 42/43 | 40/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Sulfasalazine (N=43) | Arm II: Placebo (N=42)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tenesmus (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Sulfasalazine (N=43) | Arm II: Placebo (N=42)
Anemia (Blood and lymphatic system disorders) | 15 (53) | 17 (82)
Sick sinus syndrome (Cardiac disorders) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 15 (56) | 22 (68)
Anal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 15 (40) | 15 (57)
Diarrhea (Gastrointestinal disorders) | 33 (150) | 32 (154)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 17 (44) | 15 (40)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (5) | 2 (2)
Rectal pain (Gastrointestinal disorders) | 2 (6) | 0 (0)
Tenesmus (Gastrointestinal disorders) | 17 (43) | 16 (49)
Fatigue (General disorders) | 3 (9) | 2 (6)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 1 (2) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 1 (2)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 1 (3)
Lymphocyte count decreased (Investigations) | 2 (2) | 7 (33)
Neutrophil count decreased (Investigations) | 4 (5) | 6 (14)
Platelet count decreased (Investigations) | 4 (11) | 8 (15)
White blood cell decreased (Investigations) | 8 (22) | 18 (57)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (5)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (5)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (2) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less